CLINICAL TRIAL: NCT03001570
Title: Accelerated Modulated Fractionation (SIB-IMRT) for the Treatment of Locally Advanced Squamous Cell Carcinoma From Head and Neck District
Brief Title: Accelerated Modulated Fractionation (SIB-IMRT) for Head and Neck District
Acronym: FAMOSO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: European Institute of Oncology
Record Dates: First submitted 2016-12-12; First posted 2016-12-23 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma of the Head and Neck
MeSH Terms: interventions — Cetuximab; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Radiotherapy treatment associated with concurrent Cetuximab administration.
  Patients candidate to curative concurrent Cetuximab and Radiotherapy are eligible for this study. After expressing written informed consent, patients will perform CT simulation. Then an IMRT-SIB (Simultaneous Integrated Boost) treatment plan will be elaborated and deliver the following Cetuximab pharmacokinetic:
  Length: 6 weeks; 1 fraction daily (From Monday to Friday) 30 Total Fractions (5 per week, 6 weeks of treatment). Cetuximab will be administered weekly from a week before starting radiotherapy until the end of treatment for 7 subsequent administration accordingly to the standard schedule (1 before and 6 during radiotherapy).
  Interventions: Drug: Cetuximab plus Radiotherapy

INTERVENTIONS:
Drug: Cetuximab plus Radiotherapy — Standard dose of a curative radiotherapy treatment is 70Gy given with conventional fractionation (2G daily) in an overall length of 7 weeks. In this study, the fractionation has been modified accordingly Cetuximab pharmacokinetics. Cetuximab will be administered with standard schedule: charge dose of 400mg/mq a week before the beginning of concurrent treatment, then weekly doses of 250mg/mq intravenous for 7 administration. This schedule to obtain the same biological efficacy on tumour with lower toxicity on healthy tissues.
  Other Names: Radiotherapy, IMRT

SUMMARY:
Nowadays the association between radiotherapy and the anti- Epidermal Growth Factor Receptor (anti-EGFR) monoclonal antibody Cetuximab represents a valid option in the treatment of head and neck locally advanced squamous neoplasm and, particularly, of oropharynx carcinoma. Up to date we have only indirect comparison with the standard curative treatment (i.e. concurrent radiochemotherapy) and the preliminary data show equivalent efficacy of both regimens. For this reason, concurrent Cetuximab and radiotherapy is administered in patients not eligible to chemoradiotherapy. The introduction of Cetuximab has been associated to new kind of toxicities, especially cutaneous, that have increasingly reported.

The aim of our study is to improve the toxicity/benefit ratio in patients receiving concurrent radiotherapy and cetuximab for locally advanced head and neck neoplasm. Hence, this improvement could be achieved by modulating radiation therapy dose per fraction following Cetuximab pharmacokinetics.

DETAILED DESCRIPTION:
Radiobiological rationale Overexpression of EGFR has been found to be involved into two different mechanisms of response to ionizing radiations: the former is related to the increased cell proliferation rate, the latter leading to lower radiosensitivity.

1. Increasing of cell proliferation rate From an analysis of the already reported evidences, we quantified the effect of a higher cell proliferation rate due to overexpression of EGFR. These findings were reported in patients affected with squamous carcinoma of head and neck district and evaluated for EGFR status. In those patients, local recurrence was compared in patients with different length of treatment but at the same fractionation. Consequently, the real doubling time in the subgroups with high and low EGFR expression was extrapolated . From these extrapolated values, equivalent doses of each day of non-delivered treatment have been calculated for patients who received accelerated schedule. Furthermore, doses were reported in relation to the different primary sites (oropharynx, larynx, oral cavity, hypopharynx).

   Modification of doubling time (TD) of neoplastic cell population in patients with Low and High EGFR expression.
2. Reduction of radiosensitivity Unfortunately, how radiosensitizing drugs can modify radiosensitivity cannot be evaluated retrospectively. Actually, the efficacy is evaluated on the basis of an overall effect of the treatment but radiosensitivity changes day by day in radiation and pharmacological concurrent treatment. However, these changing in radiosensitivity can be analysed in pre-clinical setting. In many reports, a progressively higher radiosensitivity has been shown in cellular survival curves by increasing EGFR inhibitor concentration. Nevertheless, the concentrations of EGFR inhibitor do not correspond to in vivo concentration during radiotherapy delivery. Fortunately, this data is obtainable from Cetuximab pharmacokinetic curve. Therefore, cell survival curves corresponding to drug concentration were obtained by performing a graphic interpolation. From these curves, daily radiosensitivity parameters were found.

Subsequently, daily doses with respect to daily radiosensitivity were identified by radiobiological calculation model. This fractionation, designed on Cetuximab pharmacokinetics, have been calculated to be equivalent to curative treatment (70Gy given with conventional schedule).

At the same time, lower cutaneous toxicity is expected with this "modulated" schedule due to the possibly increased cellular repair. Pharmacokinetics data of Cetuximab we found on the population: Vmax 4.38mg/h (15.4%), Km 74g/ml, central compartment volume Vl 2.83 l (18.6%), peripheral compartment volume 2.43 l (56.4%) and intercompartmental clearance 0.103 l/h (97.2%). Those parameters remain unmodified also during prolonged therapies. Administrated doses have been found to be adequate to cell wall receptors saturation.

A definition of overexpression of EGFR is still lacking. Different cut-offs have been proposed to distinguish patients with "high expression" from patients with "low expression" of EGFR. In a recent study the adoption of accelerated fractionation showed an advantage for those patients with an expression of EGFR>50%. Thus, we adopted this cut-off in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proof of locally advanced squamous carcinoma of oropharynx, larynx, hypopharynx (stage III and Iva)
* Overexpression of EGFR (>50%)
* Patients previously considered non-eligible for curative radio-chemotherapy for clinical reasons.
* Performance Status (ECOG) ≤ 2
* Age ≥ 18 years
* Possibility of correct administration of treatment
* Written informed consent

Exclusion Criteria:

* Distant metastases
* Oral cavity or rhinopharynx neoplasm
* Need of cutaneous bolus
* Previous treatments on head and neck district
* Collagenopathies or other severe systemic disease
* Severe cardiopathies or myocardial infarction in the previous 12 months, serious hepatopathies or other diseases with heavy impact on general conditions.
* Psychiatric disorders or other conditions preventing from expressing informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experienced acute toxicity with Grade 3 or Grade 4 adverse events according to Scala CTCAE v4.0 toxicity criteria and scale Radiation Therapy Oncology Group/European Organisation for Research and Treatment of Cancer (RTOG / EORTC) | up to 7 days during RT treatment
  During radiotherapy, patients will be assessed weekly for acute toxicity using validated international scales.acute toxicity will be assessed with CTCAE V 4.03 (Common Terminology Criteria of Adverse Events Version 4.03) scale.
  Furthermore pain (NRS pain scale) nutritional assessment (weight in kilograms ) will be performed.

SECONDARY OUTCOMES:
Number of patients who experienced late toxicity with Grade 3 or Grade 4 adverse events according to Scala CTCAE v4.0 toxicity criteria and scale RTOG / EORTC | up to 6-8 weeks after treatment completion and then up to 2 years
  Patients will be assessed weekly for late toxicity using validated international scales.acute toxicity will be assessed with CTCAE V 4.03 (Common Terminology Criteria of Adverse Events Version 4.03) scale.
Number of patients who experienced local or distance recurrence of disease assessed through clinical and radiological controls | up to 6-8 weeks after treatment completion and then up to 2 years
  Clinical assessment will be performed through:
  1. Otolaryngology examination and laryngoscopy
     Radiological assessment will be performed through:
  2. Facial skeleton and neck MRI with and without contrast or CT with and without contrast if MRI is unfeasible.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Orecchia, Prof, Study Director — European Institute of Oncology
Locations (1):
- Division of Radiotherapy European Institute of Oncology, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No